CLINICAL TRIAL: NCT00552695
Title: Phase II Study of Lidoderm Patches Prior to Intravenous Catheter Insertion.
Brief Title: Lidocaine Patches Prior to Intravenous Insertion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Research Director, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20076689
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Need for Intravenous Catheter
Keywords: intravenous catheter; emergency department; pain
MeSH Terms: conditions — Emergencies; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lidocaine 70 mg/tetracaine 70 mg skin patch
  Interventions: Device: Lidocaine tetracaine
- 2 (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Lidocaine tetracaine — Lidocaine 70 mg/tetracaine 70 mg
  Other Names: Synera
  Arms: 1
Device: Placebo — Placebo patch identical in appearance to Synera
  Arms: 2

SUMMARY:
This study will determine whether application of a patch containing a topical anesthetic (numbing medicine) named lidocaine can reduce the pain of subsequent insertion of an intravenous catheter in Emergency Department patients.

DETAILED DESCRIPTION:
Patients will be randomly assigned to an active lidocaine patch or a patch that conatins a placebo or inactive agent. Neither the patient nor the practitioner will know which patch is used since they will appear identical.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 3,
* Need for non-emergent intravenous catheter

Exclusion Criteria:

* Unstable patients,
* Allergy to lidocaine or tetracaine

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Singer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LIDODERM Patch: Lidocaine 70 mg/tetracaine 70 mg skin patch
- Control Patch: Warm patch with no active substances
Period: Overall Study
Arm/Group | LIDODERM Patch | Control Patch
Started | 22 (August 2007) | 23 (August 2007)
Completed | 22 (September 2007) | 23 (September 2007)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIDODERM Patch | Control Patch | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 23 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.3) | 10.8 (4.5) | 10 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Secondary Outcome: Success of Intravenous (IV) Insertion
Description: Percentage of patients in whom intravenous catheter was inserted successfully
Time Frame: After first attempt of catheter insertion
Measure: Number; unit: Percentage of participants
Arm/Group | LIDODERM Patch | Control Patch
Number analyzed (Participants) | 22 | 23
Percentage of participants | 18 | 17

2. Primary Outcome: Pain on Visual Analog Scale (VAS)
Description: Pain on 100 mm Visual Aanalog Scale from 0 (no pain) to 100 (most pain).
Time Frame: 0 MINUTES
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | LIDODERM Patch | Control Patch
Number analyzed (Participants) | 22 | 23
mm | 18 [1 to 40] | 35 [20 to 59]

ADVERSE EVENTS:
Arm/Group | LIDODERM Patch | Control Patch
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No